CLINICAL TRIAL: NCT00068003
Title: Cell Harvest and Preparation for Surgery Branch Treatment Protocols
Brief Title: Harvesting Cells for Experimental Cancer Treatments
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030277; 03-C-0277; NCT00897195 (obsolete NCT alias)
Record Dates: First submitted 2003-09-04; First posted 2003-09-04 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-09-12

CONDITIONS: Melanoma; Gastrointestinal Cancer; Metastatic Cancer; Breast Cancer; Non-Small Cell Lung Cancer
Keywords: Adoptive Cell Therapy; Screening; Cell Harvest; Blood; Tumor Tissue; Natural History
MeSH Terms: conditions — Melanoma; Gastrointestinal Neoplasms; Neoplasm Metastasis; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Cancer Patients: Patients with a current diagnosis of cancer
  Interventions: Drug: Anti-CD19 CAR PBL
- 2/Healthy Volunteers: Healthy volunteers

INTERVENTIONS:
Drug: Anti-CD19 CAR PBL
  Groups: 1/Cancer Patients

SUMMARY:
Background:

The NCI Surgery Branch has developed experimental therapies that involve taking white blood cells from patients' tumor or from their blood, growing them in the laboratory in large numbers, and then giving the cells back to the patient.

Objective:

This study will collect white blood cells from normal volunteers and white blood cells and/or tumor cells, from patients who have been screened for and are eligible for a NCI Surgery Branch treatment protocol. The cells collected from normal volunteers will be used as growth factors for the cells during the period of laboratory growth. The cells and/or tumor from patients will be used to make the cell treatment product.

Eligibility:

Patients must be eligible for a NCI Surgery Branch Treatment Protocol

Normal Volunteers must meet the criteria for blood donation

Design

Both patients and normal Volunteers will undergo apheresis. Patients will then undergo further testing as required by the treatment protocol.

There is no required follow up for normal volunteers.

DETAILED DESCRIPTION:
Background:

There are numerous clinical trials underway in the National Cancer Institute Surgery Branch (NCI-SB) in which patients are administered autologous lymphocytes with anti-tumor activity generated from either peripheral blood mononuclear cells (PBMC) or tumor-infiltrating lymphocytes (TIL). All adoptive cell therapy protocols require that certain cell criteria be evaluated and met prior to enrollment.

This protocol is also designed to serve as a biorepository for samples and associated data collected on patients enrolled on NCI-SB protocols, current and historical. Patients who were enrolled prior to 2003 were not enrolled on this protocol. Their tissue and data will now be retained on this protocol for long-term storage. The protocol is concerned with the retention of serum, CSF, bone marrow, ascites fluid, PBMCs, tumor, healthy tissue samples, and CD34 purified HSCS samples collected from patients with cancer to support basic science and clinical research activities of the NCI-SB at the NIH Clinical Research Center and Center for Cancer Research.

Objectives:

To obtain autologous blood, stem cells, and/or tumor tissue from patients currently with cancer for laboratory analysis and ex vivo generation of autologous anti-tumor lymphocytes for potential future enrollment on an NCI-SB adoptive cell therapy clinical trial.

To obtain allogeneic PBMC via apheresis, whole blood, or other blood products from healthy volunteers, for use in generating anti-tumor patient lymphocytes ex vivo.

To conduct genomic, proteomic, and immunologic research studies on samples collected from patients with a current diagnosis of cancer.

Eligibility:

Patients with cancer must be >= 18 years of age and meet the laboratory safety testing for infection included in all treatment trials.

Healthy volunteers for PBMC donation must meet the safety evaluation criteria established by the FDA for donation of blood products. They must also meet the strict behavioral and medical history requirements.

Healthy volunteers for whole blood donation must meet the safety evaluation criteria established by the NIH Clinical Center Department of Transfusion Medicine (DTM) Blood Bank for screening of allogeneic whole blood donors.

Design:

Once a cancer patient is determined to be a potential candidate for one of the NCI-SB clinical trials, they will undergo an apheresis and/or tumor resection for future treatment and/or research purposes. In addition, this protocol will allow for the apheresis of healthy volunteers for allogeneic PBMC or donation of whole blood for processing into serum for use in generating autologous anti-tumor lymphocytes in the laboratory, or for research purposes.

No treatments, investigational or standard therapy, will be administered on this protocol.

ELIGIBILITY:
* ELIGIBILITY CRITERIA FOR PATIENTS WITH A CURRENT DIAGNOSIS OF CANCER:

INCLUSION CRITERIA:

* Patients must have a form of cancer currently being studied in the NCI-SB.
* Patient is able to understand and willing to sign a written informed consent document.
* Age greater than or equal to 18 years.
* Clinical performance status of ECOG 0 or 1.
* Serology

  * Seronegative for HIV antibody. (The experimental treatments being evaluated depend upon an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus may be less responsive to the experimental treatment and more susceptible to its toxicities).
  * Seronegative for hepatitis B surface antigen and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Lesions which will be harvested for the generation of TIL should be accessible via standard surgical or radiological techniques and be associated with acceptable morbidity.

EXCLUSION CRITERIA:

* Active systemic infections, coagulation disorders, or other major medical illnesses of the cardiovascular, respiratory, or immune system.
* Patients who cannot give proper informed consent to the experimental therapy due to an active psychiatric disorder or inability to understand the nature of the proposed therapy and attendant risk.
* Women of child-bearing potential who are pregnant because of the potentially dangerous effects of some of the procedures (e.g., tumor biopsy or surgery for tumor resection) on the fetus.

ELIGIBILITY CRITERIA FOR HEALTHY VOLUNTEERS:

INCLUSION CRITERIA for PBMC Donors:

* Age greater than or equal to 18 years.
* Non-reactive for HBsAg, anti-HBc, anti-HCV, anti-HIV-1/2, HBV/HCV/HIV-1 NAT, anti-HTLV-I/II, anti-T. cruzi, West Nile Virus NAT,syphilis, and babesia.
* PBMC donors must meet the strict behavioral and medical history requirements as per applicable NCI-SB Apheresis Donor SOP(s).

INCLUSION CRITERIA FOR WHOLE BLOOD DONORS:

* Age greater than or equal to 18 years.
* Whole blood donors must meet the DTM inclusion criteria for allogeneic whole blood donation.

EXCLUSION CRITERIA for PBMC Donors:

* Has had babesiosis.
* Is at risk or has Creutzfeldt-Jakob Disease.
* Is on steroid therapy or any other medication or has received vaccination that might interfere with cell preparation per Principal Investigator s (PI) discretion.
* Has ongoing illness that would cause harm to the volunteer during the apheresis procedure as determined by the PI.
* Has had yellow jaundice, liver disease, or hepatitis since the age of 11.
* Has uncontrolled diabetes.
* Has a hematologic malignancy or any bleeding abnormalities.
* Has received any type of organ transplant in the past 12 months.
* Has undergone xenotransplantation at any time.
* Has received a dura mater graft.
* If female, is pregnant or has given birth within the last six weeks.
* Has had an ear or body piercing or tattoos within the past 12 months.
* Has had a blood transfusion within the past 12 months.
* Has spent time outside the United States to a restricted country.
* Has participated in any high-risk activities.

EXCLUSION CRITERIA for Whole Blood Donors:

- Whole blood donors who do not meet the DTM criteria for allogeneic whole blood donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a current diagnosis of cancer who are 18 years of age or older - Healthy volunteers who are 18 years of age or older and meet the safety evaluation criteria established by the FDA for donation of blood products, or, meet the safety evaluation criteria established by the NIH Clinical Center Department of Transfusion Medicine (DTM) Blood Bank for screening of allogeneic whole blood donors
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2003-09-08 (Actual)

PRIMARY OUTCOMES:
Generating anti-tumor patient lymphocytes ex vivo | Approximately 20 years
  Obtain allogeneic PBMC via apheresis, whole blood, or other blood products from healthy volunteers, for use in generating anti-tumor patient lymphocytes ex vivo.
To conduct genomic, proteomic, and immunologic research studies | Approximately 20 years
  Conduct genomic, proteomic, and immunologic research studies on samples collected from patients with a current diagnosis of cancer.
To obtain autologous blood, stem cells, and/or tumor tissue from patients currently with cancer | Approximately 20 years
  Obtain autologous blood, stem cells, and/or tumor tissue from patients currently with cancer for laboratory analysis and ex vivo generation of autologous anti-tumor lymphocytes for potential future enrollment on an NCI-SB adoptive cell therapy clinical trial.

SECONDARY OUTCOMES:
Repository of specimens and associated data | Approximately 20 years
  Repository for specimens and associated data obtained on patients enrolled on NCI-SB protocols who were not consented on this protocol.
Long-term storage of data and biospecimens | Approximately 20 years
  Long-term storage of data and biospecimens collected during prospective clinical trials in patients with various cancer phenotypes, to support the research activities of the NCI-SB.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. @@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Dudley ME, Wunderlich JR, Robbins PF, Yang JC, Hwu P, Schwartzentruber DJ, Topalian SL, Sherry R, Restifo NP, Hubicki AM, Robinson MR, Raffeld M, Duray P, Seipp CA, Rogers-Freezer L, Morton KE, Mavroukakis SA, White DE, Rosenberg SA. Cancer regression and autoimmunity in patients after clonal repopulation with antitumor lymphocytes. Science. 2002 Oct 25;298(5594):850-4. doi: 10.1126/science.1076514. Epub 2002 Sep 19. PMID 12242449
- [Background] Vogelstein B, Papadopoulos N, Velculescu VE, Zhou S, Diaz LA Jr, Kinzler KW. Cancer genome landscapes. Science. 2013 Mar 29;339(6127):1546-58. doi: 10.1126/science.1235122. PMID 23539594
- [Background] Robbins PF, Lu YC, El-Gamil M, Li YF, Gross C, Gartner J, Lin JC, Teer JK, Cliften P, Tycksen E, Samuels Y, Rosenberg SA. Mining exomic sequencing data to identify mutated antigens recognized by adoptively transferred tumor-reactive T cells. Nat Med. 2013 Jun;19(6):747-52. doi: 10.1038/nm.3161. Epub 2013 May 5. PMID 23644516
- [Derived] Levin N, Kim SP, Marquardt CA, Vale NR, Yu Z, Sindiri S, Gartner JJ, Parkhurst M, Krishna S, Lowery FJ, Zacharakis N, Levy L, Prickett TD, Benzine T, Ray S, Masi RV, Gasmi B, Li Y, Islam R, Bera A, Goff SL, Robbins PF, Rosenberg SA. Neoantigen-specific stimulation of tumor-infiltrating lymphocytes enables effective TCR isolation and expansion while preserving stem-like memory phenotypes. J Immunother Cancer. 2024 May 30;12(5):e008645. doi: 10.1136/jitc-2023-008645. PMID 38816232
- [Derived] White BS, Sindiri S, Hill V, Gasmi B, Nah S, Gartner JJ, Prickett TD, Li Y, Gurusamy D, Robbins P, Rosenberg SA, Leko V. Specific recognition of an FGFR2 fusion by tumor infiltrating lymphocytes from a patient with metastatic cholangiocarcinoma. J Immunother Cancer. 2023 Apr;11(4):e006303. doi: 10.1136/jitc-2022-006303. PMID 37045473
- [Derived] Zacharakis N, Huq LM, Seitter SJ, Kim SP, Gartner JJ, Sindiri S, Hill VK, Li YF, Paria BC, Ray S, Gasmi B, Lee CC, Prickett TD, Parkhurst MR, Robbins PF, Langhan MM, Shelton TE, Parikh AY, Levi ST, Hernandez JM, Hoang CD, Sherry RM, Yang JC, Feldman SA, Goff SL, Rosenberg SA. Breast Cancers Are Immunogenic: Immunologic Analyses and a Phase II Pilot Clinical Trial Using Mutation-Reactive Autologous Lymphocytes. J Clin Oncol. 2022 Jun 1;40(16):1741-1754. doi: 10.1200/JCO.21.02170. Epub 2022 Feb 1. PMID 35104158
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-C-0277.html